CLINICAL TRIAL: NCT05131724
Title: Effectiveness of Virtual Reality on Functional Mobility During Treadmill Training in Children With Cerebral Palsy: a Randomized Clinical Trial (VirtWalkCP Project)
Brief Title: Effectiveness of Virtual Reality on Functional Mobility During Treadmill Training in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Mirari Ochandorena Acha, Associate professor, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VirtWalkCP
Record Dates: First submitted 2021-11-01; First posted 2021-11-23 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy, Spastic
Keywords: "Rehabilitation"[Mesh]; "Mobility Limitation"[Mesh]; "Virtual Reality"[Mesh]
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill training (Active Comparator): The treadmill training would be 10 sessions over 2 weeks with 30 minutes for each session (5-min warm-up; 20 min gait training; 5-min cool-down). During the sessions, treadmill speed will be maintained at 60 to 80% of the maximum speed established on an exertion test. The child will walk at 60% maximum speed in the first and final five minutes and 80% in the middle 20 minutes.
  Interventions: Other: Treadmill training
- Virtual reality (Experimental): Infants in the TTVR group will perform gait training on the treadmill simultaneously with virtual reality.
  Interventions: Other: Treadmill training with virtual reality

INTERVENTIONS:
Other: Treadmill training with virtual reality — The virtual environment will be composed of obstacles, different paths, and narrow and deviated corridors. Walking through this environment will require the infant to coordinate walking behaviour and adjust the length, height, and width of steps to negotiate the obstacles on the television screen placed at the infant's eye level in front of the treadmill. The speed, orientation, size, frequency of appearance, and shape of the obstacles will be manipulated according to individual performance following a standardized protocol. The virtual system will provide visual and auditory feedback on the success or failure of the activity to enhance motor learning. In addition, the characteristics of the environment (e.g., visibility, configuration, and distractions) will be adjusted to increase the complexity of the training.
  Arms: Virtual reality
Other: Treadmill training — The RAM870A of the Medisoft treadmill will be used. Two treadmill training sessions will be held before the onset of the intervention to familiarize the children with the equipment. During these two sessions, the treadmill training and speed will be set according to the following procedures: the ground walking speed of each child will be determined through the baseline 6MWT, then the training velocity will be set at 50% of the maximum ground speed established during the 6MWT and increased gradually based on the tolerance of each child (i.e., no complaint of fatigue, heart rate not exceeding 70% of the maximum heart rate, and a lack of gait shuffling, buckling or dragging steps more than 5 seconds during walking).
  Arms: Treadmill training

SUMMARY:
Cerebral palsy (CP), which occurs as a consequence of brain damage, has multiple deficits such as a global reduction of motor cortical activity during movement execution and inadequate processing of corticospinal and somatosensory circuits. Global registers estimate that it occurs in two to three of 1.000 live births, and spasticity is the most common disorder, occurring in 80% of children with CP. Spasticity might affect both upper and lower limbs, resulting in other deficits in joint mobility, postural reactions, selective motor control, balance, and gait. This set of impairments and deficits may lead to limitations in functional ability and autonomy in the performance of daily living activities, physical fitness, quality of life, and/or ability to participate in games and sports activities compared to neurotypical peers of the same age.

Walking is considered one of the most important activities in daily life, as it is essential for activities of daily living and social participation. Children with Gross Motor Function Classification System (GMFCS) levels I, II, and III show potential for walking, and around 75% of CP children are ambulatory. However, abnormalities in neural control and muscle weakness contribute to several gait characteristics such as slow velocity, decreased stride length, increased stance phase percentage, and increased peak ankle dorsiflexion and knee flexion, and peak hip extension moments. Consequently, this gait pattern contributes to postural instability and increased fall risk in children with CP, among others.

DETAILED DESCRIPTION:
The main objective of the present study is to evaluate the effectiveness of treadmill gait training and virtual reality comparing to treadmill gait training on functional mobility in infants with spastic cerebral palsy.

The study design is a two-arm randomized clinical trial, single-center and single-blind (evaluators). The sample will be recruited at the Hospital General de Vic, and the study will be conducted at the Universitat de Vic - Universitat Central de Catalunya (UVic-UCC).

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of spastic cerebral palsy
* Motor function levels I to III according to the Gross Motor Function Classification System
* Independent walking was acquired for more than 12 months.
* Able to ambulate for at least 10 meters with or without aids.

Exclusion Criteria:

* Orthopaedic surgery on the lower limbs in the past 12 months.
* Scheduled surgery during the period of the study.
* Orthopaedic deformities with surgery indication.
* Uncontrolled seizure disorder.
* Metallic implant in the skull.
* Hearing aid.
* Have received toxic botulin injections in the past 6 months.
* Significant cognitive or visual impairment.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Functional mobility change | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks).
  The 6-Minute Walk Test (6MWT) will be performed according to the recommendations. The test will be performed once in a 10m course layout. Participants will receive standardized instructions and encouragement. The test-retest interclass correlation coefficient of this test is 0.98. The estimated time to perform the test is 10 minutes.

SECONDARY OUTCOMES:
Static balance | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The evaluation of static balance will be performed on a stabilometric platform (SystemTM SD - Biodex), which allows stabilometric analysis based on oscillations of the centre of pressure. The children will be instructed to remain standing on the platform barefoot, with arms alongside the body, gazed fixed on a point that will appear on the platform's integrated screen (at eye level, adjusted for each child), with the base of the foot free and heels aligned. The platform also has support rails if the participant loses balance during the test and needs to hold on. Readings will be taken for 30 seconds in two conditions (eyes open and eyes closed). Displacement will be measured from the oscillations of the centre of pressure in the X (anterior-posterior) and Y (medial-lateral) axes in both conditions. The test is estimated to last 5 minutes.
Dynamic balance | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The outcome will be assessed by the Beg Balance Scale will be evaluated the dynamic or functional balance. This simple 14-item measure addresses the performance of functional balance common to daily living. Each item has a five-option scale ranging from 0 to 4 points, with a maximum overall score of 56. The points are based on the time in which a position is maintained, the distance an upper limb is able to reach in front of the body, and the time needed to complete the task. The inter-rater reliability is 0.99, demonstrating the excellent reliability of this instrument. The total execution time is approximately 20 minutes.
Walking speed | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The outcome will be assessed by the 10 Meter Walk Test (10MWT), which has excellent measurement properties and is a task-specific objective measure of stepping or walking speed within an indoor environment. The test can be completed with or without a gait trainer and is not diagnostic specific. Infants will be instructed to walk 14 meters, and their speed will be measured for 10 meters to exclude acceleration at the beginning of the gait and deceleration at the end of the gait. Physical facilitation for one step will be provided for children who cannot initiate steps within a 30-second time frame. A maximum time of 10 minutes will be provided to complete the 10m. A change of 0.1 m/s will be considered to be clinically meaningful. The inter-rater reliability of this instrument is very high, between 0.89 and 1.00(64). The total execution time is approximately 10 minutes.
Gross motor function | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The outcome will be assessed by the gross motor function measure-item set (GMFM-IS). This tool is an updated version of GMFM-66 and is considered accurate, time-efficient, and suitable for research. This scale allows quantifying the infants' gross motor function in different positions (lying down and rolling; sitting; crawling and kneeling; standing; walking, running, and jumping), scoring each item from 0 to 3 points, with higher scores denoting a better performance. Clinically meaningful change for the GMFM in children with CP aged 1.5-7 years old is 1.23 for individuals classified as GMFCS level III. The test is estimated to last 10 minutes.
Functional independence | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The outcome will be assessed by the Functional Independence Measure for Children (WeeFIM), which has excellent measurement properties to measure consistent performance of activities of daily living, functional independence, and burden of care in children with disabilities. It is a semi-structured interview that is guided by a specific manual to determine the level of assistance required for (1) self-care, (2) transfers and mobility, (3) cognition and communication. A total of 18 items are scored on a scale of 1 (indicating total assistance required for completion of the task) to 7 (complete independence), giving a total score out of a possible 126. The WeeFIM will be completed by the parents or guardians of each child.
Health-related quality of life | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The outcome will be assessed using the Pediatric Quality of Life Inventory (PedsQoL). The 23-item scale encompasses: 1) Physical Functioning (8 items), 2) Emotional Functioning (5 items), 3) Social Functioning (5 items), and 4) School Functioning (5 items), and will be completed by the parents or guardian of each child. The instructions ask how much of a problem each item has been during the past 1 month. A 5-point response scale is utilized (0= never a problem; 1= almost never a problem; 2= sometimes a problem; 3= often a problem; 4= almost always a problem).
Occupational participation | Basal assessment, at the end of the intervention (an average of 3 weeks), 1 month after the end of the intervention (an average of 8 weeks)
  The outcome will be assessed using the Children Participation Questionnaire (CPQ). This questionnaire will be completed by the parents or guardians of each child. It documents the child's participation in 6 occupational areas: 1) activities of daily living; 2) instrumental activities; 3) play; 4) leisure; 5) social participation; and 6) education. Parents will report the intensity of the level of independence and the infant's enjoyment and satisfaction. It consists of 44 items that are scored on a 6-point scale (1 - 6). A higher score is considered as higher enjoyment or satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mirari Ochandorena-Acha, PhD, Principal Investigator — University of Vic - Central University of Catalonia
Locations (1):
- Univeristy of Vic - Central University of Catalonia, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication

REFERENCES:
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Chiu HC, Ada L, Bania TA. Mechanically assisted walking training for walking, participation, and quality of life in children with cerebral palsy. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD013114. doi: 10.1002/14651858.CD013114.pub2. PMID 33202482
- [Background] Grecco LAC, Hugo P, Sampaio LMM, Oliveira CS. Evidence of the effect of treadmill training on children with cerebral palsy: A systematic review. Clin Exp Med Lett [Internet]. 2012;53(2):95-100. Available from: http://www.ceml-online.com/fulltxt.php?ICID=883582
- [Background] Grecco LA, Tomita SM, Christovao TC, Pasini H, Sampaio LM, Oliveira CS. Effect of treadmill gait training on static and functional balance in children with cerebral palsy: a randomized controlled trial. Braz J Phys Ther. 2013 Jan-Feb;17(1):17-23. doi: 10.1590/s1413-35552012005000066. PMID 23538455
- [Derived] Ochandorena-Acha M, Terradas-Monllor M, Nunes Cabrera TF, Torrabias Rodas M, Grau S. Effectiveness of virtual reality on functional mobility during treadmill training in children with cerebral palsy: a single-blind, two-arm parallel group randomised clinical trial (VirtWalkCP Project). BMJ Open. 2022 Nov 3;12(11):e061988. doi: 10.1136/bmjopen-2022-061988. PMID 36328390